CLINICAL TRIAL: NCT06398730
Title: A Phase 1, Single-Center, Open-Label, Single-Arm, Dose-Escalation, Positron Emission Tomography Study to Assess the Safety and Tolerability, Immunogenicity, Pharmacokinetics, Dosimetry and Biodistribution Following GEH200521 (18F) Injection Co-Administered With GEH200520 Injection in Healthy Volunteers
Brief Title: A Phase 1, Dose-Escalation, Positron Emission Tomography Study to Assess the Safety, Pharmacokinetics, Dosimetry and Biodistribution of GEH200521 (18F) Injection Co-Administered With GEH200520 Injection in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: PPD Development, LP (Industry); Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-269-004
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- A non-radiolabeled GEH200520 - 1 mg (Experimental)
  Interventions: Drug: GEH200520 Injection and GEH200521 (18F) Injection; Diagnostic Test: Static - PET/CT scan
- A non-radiolabeled GEH200520 - 2 mg (Experimental)
  Interventions: Drug: GEH200520 Injection and GEH200521 (18F) Injection; Diagnostic Test: Static - PET/CT scan
- A non-radiolabeled GEH200520 - 4 mg (Experimental)
  Interventions: Drug: GEH200520 Injection and GEH200521 (18F) Injection; Diagnostic Test: Static - PET/CT scan
- A non-radiolabeled GEH200520 - 6 mg (Experimental)
  Interventions: Drug: GEH200520 Injection and GEH200521 (18F) Injection; Diagnostic Test: Static - PET/CT scan
- A non-radiolabeled GEH200520 - 8 mg (Experimental)
  Interventions: Drug: GEH200520 Injection and GEH200521 (18F) Injection; Diagnostic Test: Static - PET/CT scan
- A non-radiolabeled GEH200520 - 10 mg (Experimental)
  Interventions: Drug: GEH200520 Injection and GEH200521 (18F) Injection; Diagnostic Test: Static - PET/CT scan
- A non-radiolabeled GEH200520 - 12 mg or 15 mg (Experimental)
  Interventions: Drug: GEH200520 Injection and GEH200521 (18F) Injection; Diagnostic Test: Static - PET/CT scan

INTERVENTIONS:
Drug: GEH200520 Injection and GEH200521 (18F) Injection — Administration of GEH200520 Injection followed by GEH200521 (18F) Injection
Diagnostic Test: Static - PET/CT scan — Repeat whole body static scan starting 3 minutes after injection followed by a single whole body static scan at 2 to 3 hours after injection and 4 to 5 hours after injection

SUMMARY:
This is a Phase 1, single-center, open-label, single-arm, dose-escalation positron emission tomography study to assess the safety and tolerability, immunogenicity, Pharmacokinetics, dosimetry, and biodistribution after GEH200521 (18F) Injection is co-administered with GEH200520 Injection in healthy volunteers.

The estimated study duration for each subject is approximately 28 days in part A and 34 days in part B.

The primary study objective is to evaluate the safety and tolerability of the IMPs, the selected mass doses of GEH200520 Injection co-administered with a fixed dose of GEH200521 (18F) Injection.

ELIGIBILITY:
Inclusion Criteria:

* The subject is able and willing to comply with all study procedures as described in the protocol, and has read, signed, and dated an informed consent form prior to any study procedures being performed.
* The subject is male or female ≥18 years of age.
* The subject has a body mass index (BMI) ≥18 and ≤35 kg/m2.
* The subject has no history of chronic medical illness or symptoms of active illness per Investigator's assessment.
* The subject has no clinically significant deviation from normal ranges in physical examination, ECG, and clinical laboratory parameters.
* Female and male contraception methods.

Exclusion Criteria:

* Subject is using prescribed and/or non-prescribed medication which in the Investigator's opinion might impact subject safety or the study results.
* Subject has a known or suspected allergy to IMP and/or IMP ingredients.
* Subject has had a surgery within 8 weeks prior to enrollment or a surgery is scheduled during the study.
* Subject has been enrolled in this or another interventional clinical study within the 30 days before screening for this study or is actively participating in another clinical study with IMP(s).
* Subject has been enrolled in another clinical study with radiation or exposed to radiation due to medical practice, which in the Investigator's opinion might impact subject safety or the study results.
* Subject is pregnant, planning to become pregnant, or is lactating.
* Creatinine and liver function laboratory values higher than 1.5x upper limit ranges per local site clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of all TEAEs | 7 days
  Incidence of all grading of TEAEs per National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 based on the causality to the IMPs.

SECONDARY OUTCOMES:
Radiation dosimetry and biodistribution of GEH200521 (18F) Injection after the GEH200520 Injection mass doses. | 7 days
Optimal imaging window post-GEH200521 (18F) Injection after the GEH200520 Injection mass doses. | 7 days
Mass dose of GEH200520 Injection followed by a fixed dose of GEH200521 (18F) Injection to achieve a diagnostic positron emission tomography (PET) image quality. | 7 days
Pharmacokinetic property of the area under the curve (AUC) of total protein following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection. | 7 days
Pharmacokinetic property of Cmax of total protein following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection. | 7 days
Pharmacokinetic property of clearance (CL) of total protein following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection. | 7 days
Pharmacokinetic property volume of distribution (V) of total protein following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection. | 7 days
To characterise the pharmacokinetic property of the elimination half-life (t1/2) of total protein following administration of different GEH200520 Injection mass doses with a fixed dose of GEH200521 (18F) Injection. | 7 days
Collection of the incidence, severity, changes between visits for AEs/SAEs/AESIs. | 7 days
Proportion of subjects with clinically significant abnormalities detected during physical examination status by system organs following administration of GEH200520 and GEH200521 (18F). | 7 days
Proportion of subjects with clinically significant abnormalities detected for serum biochemistry test results following administration of GEH200520 and GEH200521 (18F). | 7 days
Proportion of subjects with clinically significant abnormalities detected for haematology test results following administration of GEH200520 and GEH200521 (18F). | 7 days
Proportion of subjects with clinically significant abnormalities detected for beats per minute following administration of GEH200520 and GEH200521 (18F). | 7 days
Changes in systolic and diastolic blood pressure in mmHg following administration of GEH200520 and GEH200521 (18F). | 7 days
Changes in temperature as degree F following administration of GEH200520 and GEH200521 (18F). | 7 days
Proportion of subjects with clinically significant abnormalities detected during 12-lead electrocardiograms (ECGs) following administration of GEH200520 and GEH200521 (18F). | 7 days
Incidence of treatment induced and treatment enhance anti drug antibody responses following administration of GEH200520 and GEH200521 (18F) | 7 days
Test-retest imaging reliability of GEH200521 (18F) Injection co-administered with the selected mass dose of GEH200520 Injection, when administered on 2 different days | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Raiter, Study Director — GE Healthcare
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No